CLINICAL TRIAL: NCT02512341
Title: Automatic Differentiation of Innocent and Pathologic Murmurs in Pediatrics
Status: Completed | Type: Observational
Sponsor: CSD Labs GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: OTT01
Record Dates: First submitted 2015-07-29; First posted 2015-07-30 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Heart Murmurs; Mitral Valve Prolapse; Systolic Murmurs
Keywords: Computer Aided Auscultation (CAA); Electronic Stethoscope; Phonocardiography; Heart Auscultation
MeSH Terms: conditions — Heart Murmurs; Mitral Valve Prolapse; Systolic Murmurs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Computer Aided Auscultation (CAA)
  Other Names: Phonocardiogram analysis; Automated heart murmur classification; Murmur screening

SUMMARY:
The purpose of this preliminary clinical study is to assess the quality of a computational algorithm that automatically classifies murmurs of phonocardiograms (PCGs) as either pathologic (AHA class I) or as no- or innocent (AHA class III) in the pediatric population.

Each patient is auscultated and diagnosed independently by a medical specialist by means of a standard mechanical stethoscope. Additionally, for each patient, a PCG is recorded using a Littmann 3200 electronic stethoscope and later analyzed using the computational algorithm. An echocardiogram is performed as the gold-standard for determining heart pathologies. The results of the computer aided auscultation (CAA) are compared to the findings of the medical professionals as well as to the echocardiogram findings.

Hypothesis: The specific CAA algorithms used in this study are able to differentiate pathologic (AHA class I) from no- or innocent murmurs (AHA class III) in a pediatric population.

DETAILED DESCRIPTION:
Background:

Computer aided auscultation in the differentiation of pathologic (AHA class I) from no- or innocent murmurs (AHA class III) would be of great value to the general practitioner and potentially also to the specialist. This would allow objective screening for structural heart disease, standardized documentation of auscultation findings, and may avoid unnecessary referrals to pediatric cardiologists. Our goal was to further develop and assess the quality of a novel computational algorithm that automatically classifies murmurs of phonocardiograms (PCGs) acquired in a pediatric population.

Methods:

Patients with no-, innocent-, and pathologic murmurs were recruited from the general pediatric cardiology clinic. Using an electronic stethoscope, PCGs were acquired by the pediatric cardiologist from each patient. The PCGs were analyzed by the algorithm and diagnoses were compared to findings by the pediatric specialist and echocardiography as the gold standard.

The following registry procedures and quality factors have been implemented in this preliminary clinical study:

* Quality assurance plan, including

  * data validation
  * proper registration procedures
* Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources (medical records and paper case report forms).
* Standard Operating Procedures to address registry operations and analysis activities, including patient recruitment, data collection, data management, data analysis.

ELIGIBILITY:
Inclusion Criteria:

* outpatient
* parental approval for study participation

Exclusion Criteria:

* none

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Outpatients with and without heart defects showing pathological heart murmurs, innocent heart murmurs and heart sounds without murmurs at the cardiology department.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of correctly diagnosed pathological heart murmurs through independent algorithm-based auscultation. | 2 months
  Each patient is screened and diagnosed regarding a potential heart murmur by a medical expert through standard stethoscope-based auscultation. Heart sounds are recorded using an electronic Littmann 3200 stethoscope. The resulting phonocardiograms are analyzed and diagnosed independently, offline, with no external input, by an algorithm. A final diagnosis for each patient is made by a medical expert by performing an echocardiogram, the gold standard method for heart murmur detection. The diagnoses of both the medical expert and the algorithm are finally compared to the echocardiogram-based diagnosis.

SECONDARY OUTCOMES:
Number of correctly diagnosed pathological heart murmurs through traditional stethoscope based auscultation by medical experts. | 2 months
  Each patient is screened and diagnosed regarding a potential heart murmur by a medical expert through standard stethoscope-based auscultation. Heart sounds are recorded using an electronic Littmann 3200 stethoscope. The resulting phonocardiograms are analyzed and diagnosed independently, offline, with no external input, by an algorithm. A final diagnosis for each patient is made by a medical expert by performing an echocardiogram, the gold standard method for heart murmur detection. The diagnoses of both the medical expert and the algorithm are finally compared to the echocardiogram-based diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Lai, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Canada